CLINICAL TRIAL: NCT06911450
Title: Quantification of Pleural Longitudinal Strain by Speckle-Tracking Ultrasound: Feasibility and Associations With Driving Pressure in Mechanically Ventilated Patients
Brief Title: Pleural Strain by Speckle-Tracking Ultrasound: Feasibility and Driving Pressure Associations
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Pleural Strain by Speckle-Tracking Ultrasound and Driving Pressure in Ventilated Patients, First Affiliated Hospital of Wannan Medical College
Other Study IDs: 2024174
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Ventilation, Mechanical; ARDS (Acute Respiratory Distress Syndrome)
Keywords: Speckle-Tracking Ultrasound; Pleural Longitudinal Strain; Mechanical Ventilation; Ventilator-Induced Lung Injury (VILI); Lung Strain
MeSH Terms: conditions — Respiratory Aspiration; Acute Lung Injury; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Phase one: This phase aims to evaluate the feasibility and consistency of speckle-tracking technology for measuring pleural longitudinal strain. A cohort of 25 critically ill non-ventilated patients (APACHE II score >8) was enrolled. A single operator acquired 10-second pleural videos at the upper blue point position using a GE Vivid iq ultrasound system (GE Healthcare, USA) with a superficial probe. Two independent operators subsequently analyzed the lung ultrasound (LUS) clips offline using GE EchoPAC software (version 203, GE Healthcare, USA) to derive the maximum pleural longitudinal strain. Each measurement was performed three times, and the average value was recorded. The same measurements were repeated one week later. Inter- and intra-observer consistency was assessed using the intraclass correlation coefficient (ICC), where values range from 0 (poor agreement) to 1 (perfect agreement). An ICC >0.75 was predefined as indicating good consistency, thereby validating the feasibility of apply
- Phase two: This phase evaluates the feasibility and reproducibility of speckle-tracking technology in mechanically ventilated patients. Twenty-five eligible mechanically ventilated patients were included. Ultrasound acquisition and pleural strain measurement protocols mirrored those in Phase 1. To assess intra-operator reproducibility, each operator performed duplicate measurements at 10-minute intervals. Operators were blinded to each other's results, and each parameter was measured three times with the average value recorded. Inter- and intra-observer consistency was analyzed using ICC, with thresholds identical to Phase 1 (ICC >0.75 indicating acceptable reproducibility).
- Phase three: This phase investigates the correlation between pleural longitudinal strain and driving pressure (ΔP) in 25 mechanically ventilated patients. Speckle-tracking ultrasound was used to measure pleural strain at three distinct driving pressure levels (10, 15, and 20 cmH₂O). The Pearson correlation coefficient was employed to quantify the linear relationship between pleural strain (continuous variable) and driving pressure. Statistical significance was defined as a two-tailed p-value <0.05.

SUMMARY:
What is this study about? This research aims to test a new ultrasound technology called "speckle tracking" to measure how much the lining of your lungs (pleura) stretches during breathing, especially if you're on a breathing machine (ventilator). Doctors want to see if this technology can help them adjust ventilator settings more safely, reducing the risk of lung damage.

Why is this important? Lung protection: Patients on ventilators, especially those with severe lung problems (like ARDS or pneumonia), need careful settings. Too much pressure from the ventilator can harm the lungs.

Better monitoring: Current tools can't easily measure lung stretching at the bedside. This ultrasound method might offer a simple, painless way to check lung health in real time.

Who can join? Included: Adults (18+ years) in the ICU with serious illness (assessed by a standard score called APACHE II >8), whether on a ventilator or not.

Excluded: People with recent chest surgery, broken ribs, nerve/muscle diseases, or pregnancy (to avoid risks and ensure accurate measurements).

What will happen during the study?

Ultrasound scans:

A small probe will be placed gently on your chest for 5-10 minutes. The machine will record videos of your lung movements during breathing. This is painless and uses no radiation.

Measurements:

Doctors will repeat the scan twice (10 minutes apart) to check consistency. For ventilator patients, scans will be done at different pressure settings to see how lung stretching changes.

How will this help me or others? Direct benefit: You'll receive detailed monitoring of your lung function, which may help doctors personalize your care.

Future benefit: If successful, this technology could help doctors worldwide adjust ventilators more safely, reducing complications for ICU patients.

Is my information safe? All data (scans, medical records) will be anonymized and stored securely. Participation is voluntary, and you can withdraw anytime without affecting your treatment.

Who is conducting the study? Led by Dr. Xu Qiancheng and the ICU team at Yijishan Hospital, Wannan Medical College.

Experts in ultrasound and critical care will ensure the study is safe and scientifically rigorous.

ELIGIBILITY:
Phase 1: Feasibility Assessment in Non-Mechanically Ventilated Patients

Inclusion Criteria:

* Adult patients (≥18 years) admitted to the ICU with an APACHE II score >8.
* Non-mechanically ventilated patients (either spontaneously breathing or receiving only non-invasive oxygen therapy).

Exclusion Criteria:

* History of thoracic surgery or trauma.
* Presence of pneumothorax or chest trauma (e.g., rib fractures, flail chest).
* Pregnancy or age <18 years.
* Refusal to participate by the patient or legal representative.
* Poor ultrasound image quality (e.g., unclear pleural visualization).

Phase 2: Feasibility Assessment in Mechanically Ventilated Patients

Inclusion Criteria:

* Adult patients (≥18 years) admitted to the ICU with an APACHE II score >8.
* Receiving invasive mechanical ventilation for >24 hours.

Exclusion Criteria:

* History of thoracic surgery or trauma.
* Presence of pneumothorax or chest trauma (e.g., rib fractures, flail chest).
* Pregnancy or age <18 years.
* Requirement for high-frequency oscillatory ventilation.
* Poor ultrasound image quality (e.g., pleural motion obscured by pleural effusion).

Phase 3: Correlation Analysis of Strain and Driving Pressure in Mechanically Ventilated Patients

Inclusion Criteria:

* Adult patients (≥18 years) admitted to the ICU with an APACHE II score >8.
* Receiving invasive mechanical ventilation for >24 hours.
* Tolerance to stepwise driving pressure adjustments (10, 15, and 20 cmH₂O, maintained for 10 minutes each).

Exclusion Criteria:

* History of thoracic surgery or trauma.
* Presence of pneumothorax, chest trauma (e.g., rib fractures, flail chest), or significant patient-ventilator asynchrony.
* Pregnancy or age <18 years.
* Requirement for high-frequency oscillatory ventilation.
* Hemodynamic instability (mean arterial pressure [MAP] <65 mmHg or requiring high-dose vasopressors).
* Severe hypoxemia (PaO₂/FiO₂ <100 mmHg), precluding safe adjustment of driving pressure.
* Poor ultrasound image quality (e.g., loss of pleural strain signal).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study enrolls critically ill patients in the intensive care unit (ICU) to evaluate the feasibility and clinical relevance of speckle-tracking ultrasound for pleural strain measurement. The study population is divided into three sequential phases:
  Phase 1 Cohort:
  25 non-ventilated patients (spontaneously breathing or on non-invasive oxygen therapy) with an APACHE II score >8.
  Focus: Technical validation of pleural strain measurement feasibility.
  Phase 2 Cohort:
  25 mechanically ventilated patients (invasive ventilation >24 hours) with an APACHE II score >8.
  Focus: Reproducibility of strain measurement under ventilator-induced motion artifacts.
  Phase 3 Subgroup:
  A subset of 25 patients who tolerate driving pressure adjustments (10, 15, 20 cmH₂O).
  Focus: Correlation between pleural strain and driving pressure.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of speckle-tracking ultrasound for pleural longitudinal strain measurement | At baseline (Day 1)
  The feasibility is defined as achieving inter- and intra-observer consistency with an intraclass correlation coefficient (ICC) >0.75.
  Measurement: ICC calculated from three repeated strain measurements by two independent operators.
  Threshold: ICC >0.75 indicates acceptable feasibility.
Correlation between pleural longitudinal strain and driving pressure | During ventilator adjustment (Day 1)
  The strength of the linear relationship between pleural strain (continuous variable) and driving pressure (ΔP) measured by Pearson's correlation coefficient.
  Threshold: A Pearson's r >0.5 with a p-value <0.05 is predefined as a clinically significant correlation.

SECONDARY OUTCOMES:
Time required for ultrasound analysis | Immediately post-procedure (Day 1)
  Total time (minutes) to acquire and analyze pleural strain data, reported as mean ± SD.
Success rate of pleural strain measurement | At baseline (Day 1)
  Percentage of patients with analyzable pleural strain data (e.g., clear speckle-tracking signal).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes